CLINICAL TRIAL: NCT00184002
Title: A Phase II Study Of Pegylated Liposomal Doxorubicin (Doxil) In Combination With Rituxan, Cyclophosphamide, Vincristine and Prednisone (DR-COP) In Newly Diagnosed Aggressive Non-Hodgkin's Lymphomas
Brief Title: Doxorubicin (Doxil) Combined With Rituxan, Cyclophosphamide, Vincristine and Prednisone in Newly Diagnosed Aggressive Non-Hodgkin's Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13NHL-02-3
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Doxorubicin; Rituximab; Cyclophosphamide; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DR-COP (Experimental): On cycle 1 patients receive Doxil 40 mg/m2 iv day 1 over a minimum of 60 min., Cyclophosphamide 750 mg/m2 iv day 1 over a minimum of 60 min., Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum) and Prednisone 100 mg po days 1-5.
  On cycle 2 until study completion patients receive Doxil 40 mg/m2 iv day 1, Rituxan 375 mg/m2 iv day 1, Cyclophosphamide 750 mg/m2 iv day 1, Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum) and Prednisone 100 mg po days 1-5
  * 1 cycle = 21 days.
  * Continue treatment until 2 cycles beyond documentation of CR for a maximum of 8 cycles.
  Interventions: Drug: Doxorubicin, Rituxan, Cyclophosphamide, Vincristine and Prednisone

INTERVENTIONS:
Drug: Doxorubicin, Rituxan, Cyclophosphamide, Vincristine and Prednisone — Cycle 1 Doxil 40 mg/m2 iv day 1 over a minimum of 60 min.
  Cyclophosphamide 750 mg/m2 iv day 1 over a minimum of 60 min.
  Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum).
  Prednisone 100 mg po days 1-5.
  Cycle 2 until study completion
  Doxil 40 mg/m2 iv day 1
  Rituxan 375 mg/m2 iv day 1
  Cyclophosphamide 750 mg/m2 iv day 1
  Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum)
  Prednisone 100 mg po days 1-5
  * 1 cycle = 21 days.
  * Continue treatment until 2 cycles beyond documentation of CR for a maximum of 8 cycles.

SUMMARY:
The current standard treatment for non-Hodgkin's lymphoma involves drugs called cyclophosphamide, doxorubicin, vincristine, prednisone and rituxan in a regimen called "R-CHOP." Using R-CHOP therapy, complete disappearance of disease is expected in over 50% of people. One of the active drugs in the R-CHOP regimen, doxorubicin, has previously been reformulated and been placed in a fatty bubble called a liposome. The reason for placing the drug in the liposome is that there is evidence that the liposome is better taken up by tumors. This liposomally encapsulated form of doxorubicin called Doxil has shown similar or better anti-tumor against certain tumors with reduced side effects. Doxil is FDA approved for ovarian cancer. However its use in non-Hodgkin's lymphoma is still investigational. By substituting Doxil for doxorubicin in the R-CHOP regimen, it is hoped this treatment will be better at shrinking tumors and with reduced side effects. The purpose of this study is to see how well the combination of Doxil, rituximab, cyclophosphamide, vincristine and prednisone (DR-COP) are in shrinking tumors in patients with non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of Non-Hodgkin's lymphoma of B-cell origin: follicular large cell, diffuse large cell (including all B-cell variants), Burkitt or Burkitt-like lymphoma
* All stages of disease
* Measurable or evaluable tumor parameter(s)
* Age greater than 17 years old
* Karnofsky performance status greater or equal to 50%
* AGC greater or equal to 1.0; platelets greater or equal to 75,000(unless abnormal because of lymphoma)
* Bilirubin less or equal to 2.0; SGOT less or equal to 3 times upper limit of normal (unless abnormal because of lymphoma)
* Creatinine less or equal to 2.0 or creatinine clearance greater or equal to 60 ml/min (unless abnormal because of lymphoma)
* LVEF greater or equal to 45%
* Concurrent RT with or without steroids for emergency conditions secondary to lymphoma (i.e., CNS tumor, cord compression)are permitted
* Men and women of childbearing potential must agree to use adequate birth control for the duration of the therapy and for 3 months after completion of therapy
* Signed informed consent

Exclusion Criteria:

* Prior systemic cytotoxic therapy or RT for lymphoma
* Second active tumor, other than non-melanomatous skin ca and in-situ cervical cancer
* HIV seropositive
* Primary CNS lymphoma
* Pregnant or nursing women
* Unable to comply with the requirements of the protocol, or unable to provide adequate informed consent, in the opinion of the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-01-10 (Actual); Primary Completion 2012-12-19 (Actual); Study Completion 2013-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Tulpule, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study began recruiting in January 2003 and ended in December 2007. All subjects were seen and treated either at USC Norris Comprehensive Cancer Center or at LAC+USC Medical Center.
Pre-assignment Details: There were no pre-assignment criteria. All subjects were given the same treatment.
Groups:
- DR-COP: On cycle 1 patients receive Doxil 40 mg/m2 iv day 1 over a minimum of 60 min., Cyclophosphamide 750 mg/m2 iv day 1 over a minimum of 60 min., Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum) and Prednisone 100 mg po days 1-5.
  On cycle 2 until study completion patients receive Doxil 40 mg/m2 iv day 1, Rituxan 375 mg/m2 iv day 1, Cyclophosphamide 750 mg/m2 iv day 1, Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum) and Prednisone 100 mg po days 1-5
  * 1 cycle = 21 days.
  * Continue treatment until 2 cycles beyond documentation of CR for a maximum of 8 cycles.
  Doxorubicin, Rituxan, Cyclophosphamide, Vincristine and Prednisone: Cycle 1 Doxil 40 mg/m2 iv day 1 over a minimum of 60 min.
  Cyclophosphamide 750 mg/m2 iv day 1 over a minimum of 60 min.
  Vincristine 1.4 mg/m2 iv bolus day 1 (2.0 mg maximum).
  Prednisone 100 mg po days 1-5.
  Cycle 2 until study completion
  Doxil 40 mg/m2 iv day 1
  Rituxan 375 mg/m2 iv day 1
  Cyclophosphamide 750 mg/m2 iv day 1
Period: Overall Study
Arm/Group | DR-COP
Started | 68
Completed | 51
Not Completed | 17
Not completed — Adverse Event | 9
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | DR-COP
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 48
Region of Enrollment [Number; unit: participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Complete Response to the Combination Chemotherapy
Description: Initial disease response tests will be performed after cycle 4 on all patients. Subsequent assessments after cycles 6 and/or 8 will depend on response. If after 4 cycles of therapy complete response or partial response has been documented, therapy will continue. If stable or progressive disease has been documented, the patient will be withdrawn from the study.
  Response to the study treatment will be determined according to the criteria proposed in the "Report of an International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphomas" by Cheson et al (23).
Time Frame: At completion of cycle 4, 6, and 8
Measure: Number; unit: Percentage of participants
Arm/Group | DR-COP
Number analyzed (Participants) | 68
Percentage of participants
  Complete Response | 75.0
  Partial Response | 23.0

2. Secondary Outcome: Number of Patients With Serious Adverse Events as a Measure of Safety and Tolerability
Description: Summary of grade 3 or higher toxicities (per Common Toxicity Criteria version 2.0) which generally is described as severe adverse reaction or symptom.
Time Frame: At end of every cycle
Measure: Count of Participants; unit: Participants
Arm/Group | DR-COP
Number analyzed (Participants) | 68
Participants | 35

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning cycle 1 and continued throughout the study until 30 days after the last dose.
Arm/Group | DR-COP
All-Cause Mortality (participants affected / at risk) | 3/68
Serious Adverse Events (participants affected / at risk) | 35/68
Other Adverse Events (participants affected / at risk) | 27/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-COP (N=68)
Abdominal pain or cramping (Gastrointestinal disorders) | 2 (4)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 35 (42)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (Hepatobiliary disorders) | 1 (1)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Cardiac troponin I (cTnl) (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 1 (1)
Febrile neutropenia (Infections and infestations) | 8 (8) — Fever of unknown origin without clinically or microbiologically documented infection (ANC <1.0 x 10e9/L, fever >= 38.5 degrees C)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 10 (10)
Hemoglobin (Blood and lymphatic system disorders) | 11 (13)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5)
Hypertension (Cardiac disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (1)
Infection (Infections and infestations) | 8 (8) — Documented clinically or microbiologically with grade 3 or 4 neutropenia (ANC <1.0 x 10e9/L)
Infection without neutropenia (Infections and infestations) | 6 (6)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neuropathy-sensory (Nervous system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 5 (9)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 3 (3)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 3 (3)
Stomatitis/pharingitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Ureteral obstruction (Renal and urinary disorders) | 1 (1)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Weight loss (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-COP (N=68)
Abdominal pain or cramping (Gastrointestinal disorders) | 12 (14)
Alkaline phosphatase (Hepatobiliary disorders) | 1 (1)
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 24 (30)
Anorexia (Metabolism and nutrition disorders) | 16 (19)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 5 (5)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Bilirubin (Hepatobiliary disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (11)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 19 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Creatinine (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Diarrhea patients without colostomy (Gastrointestinal disorders) | 12 (16)
Dizziness/lightheadedness (Nervous system disorders) | 4 (4)
Dry eye (Eye disorders) | 1 (1)
Dyspepsia/heartburn (Gastrointestinal disorders) | 7 (7)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 5 (5)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (2)
Edema (General disorders) | 11 (16)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 22 (32)
Fever (General disorders) | 11 (12) — In the absence of neutropenia, where neutropenia is defined as AGC <1.0 x 10e9/L
Flatulence (Gastrointestinal disorders) | 1 (1)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 18 (23)
Headache (Nervous system disorders) | 14 (17)
Hemoglobin (Blood and lymphatic system disorders) | 23 (42)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhage/bleeding (Injury, poisoning and procedural complications) | 1 (1) — Without grade 3 or 4 thrombocytopenia
Hot flashes/flushes (Endocrine disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (27)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Cardiac disorders) | 5 (5)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Cardiac disorders) | 3 (3)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 9 (15)
Insomnia (Psychiatric disorders) | 15 (16)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Mood alteration-anxiety, agitation (Psychiatric disorders) | 2 (2)
Mood alteration-depression (Psychiatric disorders) | 3 (3)
Mouth dryness (Gastrointestinal disorders) | 1 (1)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 22 (37)
Neuropathy-motor (Nervous system disorders) | 1 (1)
Neuropathy-sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 19 (34)
Pain due to radiation (General disorders) | 1 (1)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 2 (4)
Pain (General disorders) | 27 (63)
Platelets (Blood and lymphatic system disorders) | 6 (14)
Pleural Effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (10)
Rigors, chills (General disorders) | 3 (3)
Sense of smell (Gastrointestinal disorders) | 2 (2)
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 5 (7)
SGPT (ALT) (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 5 (8)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 7 (10)
Skin-Laate RT Morbidity Scoring (Injury, poisoning and procedural complications) | 2 (2)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 17 (24)
Sweating (eiaphoresis) (General disorders) | 2 (2)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 14 (17)
Thrombosis/embolism (Cardiac disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (22)
Weight loss (General disorders) | 2 (2)
Wound-infectious (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes